CLINICAL TRIAL: NCT07393048
Title: Application and Exploration of Personalized ctDNA-MRD Detection Technology in Predicting the Efficacy of Neoadjuvant Therapy for Rectal Cancer
Acronym: ctDNA-MRD-RC
Status: Recruiting | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Yao Hongwei, Professor, Beijing Friendship Hospital
Other Study IDs: MR-11-26-002019
Record Dates: First submitted 2026-01-12; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Locally Advanced Rectal Cancer (LARC)
Keywords: ctDNA-MRD; Rectal Cancer; Neoadjuvant Therapy; Predicting the Efficacy; Detection Technology
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples, colorectal cancer tissue samples obtained via colonoscopy, or tissue slides (white sections)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rectal Cancer ctDNA-MRD Detection Cohort: This study is an exploratory study, with an expected enrollment of 60 patients diagnosed with stage II-III rectal cancer who are scheduled to undergo neoadjuvant therapy. The sample collection and testing procedures are as follows: Before neoadjuvant therapy: Baseline endoscopic biopsy tissue or paraffin sections:1.1 Two pieces of endoscopic biopsy tissue, approximately 2 mm in diameter, are collected and placed in tissue preservation tubes.1.2 Ten unstained tissue slides are prepared. Peripheral blood collection: 10 mL of blood is collected using cell-free DNA blood collection tubes for the following assays:① ctDNA-customized MRD high-depth sequencing;② ctDNA shallow whole-genome sequencing (sWGS) for monitoring copy number variation (CNV) profiles;③ Mitochondrial DNA (mtDNA) analysis. During neoadjuvant therapy (within 2 weeks after radiotherapy completion): Peripheral blood collection: 10 mL of blood is collected using cell-free DNA blood collection tubes for the followin
  Interventions: Diagnostic Test: Personalized ctDNA-MRD Detection

INTERVENTIONS:
Diagnostic Test: Personalized ctDNA-MRD Detection — This observational study involves collecting clinical data and biospecimens (peripheral blood and tissue samples) from participants at multiple timepoints. Personalized ctDNA-MRD detection technology, together with copy number variation and mtDNA profiling, is applied to analyze the samples. The primary goal is to predict neoadjuvant therapy efficacy by identifying biomarkers associated with key outcomes, such as tumor regression grade and pathological complete response rate. No experimental drugs or treatments are administered.

SUMMARY:
This study is a single-center, prospective, observational clinical trial enrolling patients with locally advanced rectal cancer (cT3-4aN0M0 and cT1-4aN1-2M0). By collecting tissue and blood samples at multiple timepoints, and integrating multi-omics data including ctDNA mutations, copy number variations, and mtDNA profiles, a multi-omics model will be constructed to predict the efficacy of neoadjuvant therapy for rectal cancer.

DETAILED DESCRIPTION:
This study is a single-center, prospective, observational clinical trial designed to construct and validate a multi-omics-based predictive model for neoadjuvant treatment efficacy in locally advanced rectal cancer. Patients diagnosed with locally advanced rectal cancer (cT3-4aN0M0 and cT1-4aN1-2M0) are enrolled, and tissue and blood samples are dynamically collected at multiple time points. By simultaneously analyzing plasma circulating tumor DNA (ctDNA) somatic mutations, copy number variations, and mitochondrial DNA (mtDNA), a multi-dimensional molecular biomarker system is constructed.The primary objectives of the study include: first, prospectively validating the efficacy of a multi-dimensional molecular biomarker model based on ctDNA mutations, mtDNA, and copy number variations for detecting molecular residual disease (MRD) during neoadjuvant therapy and assessing its sensitivity and specificity in predicting pathological response; second, comparing the sensitivity and specificity of different omics features-ctDNA mutations, mtDNA, copy number variations, alone or in combination-in predicting treatment efficacy after surgery.The secondary objectives are: first, to construct a multi-omics model integrating ctDNA mutations, copy number variations, and mtDNA for dynamically assessing tumor burden changes during neoadjuvant therapy; second, to explore and optimize ctDNA-MRD detection technology, aiming to overcome the high sample volume requirements of traditional methods and improve the detection rate of low-abundance ctDNA.

ELIGIBILITY:
Inclusion Criteria:

* 1: Signed a written informed consent form and voluntarily participated in this study
* 2: Aged 18-75 years, regardless of sex
* 3: Histopathologically confirmed rectal adenocarcinoma
* 4: Clinical stage II-III as assessed by MRI (according to the AJCC 8th edition)
* 5: Distance from the lower tumor margin to the anal verge ≤10 cm
* 6: Surgically resectable
* 7: Able to swallow tablets normally
* 8: ECOG PS 0-1
* 9: No prior antitumor therapy for rectal cancer, including radiotherapy, chemotherapy, or surgery
* 10: Scheduled to undergo surgical treatment after completion of neoadjuvant therapy
* 11: No surgical contraindications
* 12: Normal function of major organs, including: complete blood count, blood biochemistry, and coagulation function

Exclusion Criteria:

* 1: History of allergy to monoclonal antibodies, any component of tislelizumab, or capecitabine
* 2: Prior or ongoing receipt of any tumor-directed surgery, radiotherapy, chemotherapy, targeted therapy, immunotherapy, etc
* 3: Presence of any active autoimmune disease or history of autoimmune disease
* 4: History of immunodeficiency, including a positive HIV test result, other acquired or congenital immunodeficiency disorders, or history of organ transplantation or allogeneic bone marrow transplantation
* 5: Poorly controlled cardiac clinical symptoms or diseases, including but not limited to: heart failure of NYHA class II or above, unstable angina, myocardial infarction within the past year, or clinically significant supraventricular or ventricular arrhythmia that remains poorly controlled without or despite clinical intervention
* 6: Diagnosis of another malignancy within 5 years prior to the first use of the study drug, except for malignancies with low risk of metastasis or death (5-year survival rate >90%), such as adequately treated basal cell carcinoma or squamous cell carcinoma of the skin, or carcinoma in situ of the cervix, which may be considered for inclusion
* 7: Pregnant or lactating women
* 8: Other factors, as judged by the investigator, that may lead to premature termination of the study, such as other severe diseases (including psychiatric disorders) requiring concomitant treatment, alcohol abuse, drug abuse, family or social factors, or any condition that may affect the safety or compliance of the participant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: "Enrolled subjects must be 18-75 years old, pathologically confirmed with rectal adenocarcinoma (MRI stage II-III), with a tumor inferior margin ≤10 cm, resectable via surgery, ECOG performance status 0-1, normal major organ function, no prior relevant treatment, ability to take oral medications, signed informed consent, and no surgical contraindications. Detailed eligibility criteria can be found in the study protocol." "Subjects with a history of drug allergy, prior cancer treatment, active or past autoimmune disease, immunodeficiency, severe heart disease, other malignant tumors (except low-risk ones) within the past five years, pregnancy or lactation, or other factors affecting safety and compliance will be excluded from this study. Detailed eligibility criteria can be found in the study protocol."
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) rate | Post-neoadjuvant Therapy Efficacy Assessment Time Point (within 8-12 weeks after radiotherapy completion)
  The proportion of patients confirmed to have achieved complete response after neoadjuvant therapy, as assessed by endoscopy, imaging (pelvic MRI/chest-abdominal CT), digital rectal examination, and pathological evaluation. The assessment time point corresponds to T2 (8-14 weeks after the end of neoadjuvant therapy). Complete response requires: normal mucosa on endoscopy with negative biopsy; no residual tumor on imaging; no palpable mass on digital rectal examination; and no viable tumor cells in postoperative pathology (if surgery is performed).

SECONDARY OUTCOMES:
Complete Response Rate (CR) | Post-neoadjuvant Therapy Efficacy Assessment Time Point (within 8-12 weeks after radiotherapy completion)
  The proportion of patients confirmed to have achieved complete response after neoadjuvant therapy, as assessed by endoscopy, imaging (pelvic MRI/chest-abdominal CT), digital rectal examination, and pathological evaluation. The assessment time point corresponds to T2 (8-14 weeks after the end of neoadjuvant therapy). Complete response requires: normal mucosa on endoscopy with negative biopsy; no residual tumor on imaging; no palpable mass on digital rectal examination; and no viable tumor cells in postoperative pathology (if surgery is performed).
Major Pathological Response Rate (MPR) | 1 month after surgery
  The proportion of patients with ≤10% residual tumor cells and no lymph node metastasis in postoperative pathological examination, assessed at T3 (1 month after radical resection, corresponding to the technical roadmap).
Objective Response Rate (ORR) | Post-neoadjuvant Therapy Efficacy Assessment Time Point (within 8-12 weeks after radiotherapy completion)
  The proportion of patients who achieve complete response (CR) or partial response (PR) after neoadjuvant therapy, assessed at T2 (8-14 weeks after the end of neoadjuvant therapy). Partial response is defined as a ≥30% reduction in tumor size confirmed by endoscopy and imaging, with no new lesions.
Disease-Free Survival (DFS) | Monitoring Period: Every 3 or 6 months after treatment completion, continued until 1 year.
  The time from the initiation of neoadjuvant therapy to disease recurrence (confirmed by endoscopy/imaging), metastasis, or death from any cause, with follow-up through T4 (surveillance period of 3-6 months, optional) and subsequent long-term follow-up nodes as per the technical roadmap.
Overall Survival (OS) | From the randomization date to the date of death from any cause, disease recurrence, or metastasis-whichever occurred first-assessed over the entire study period with a planned maximum follow-up of 12 months.
  Time from randomization to death from any cause, recurrence, or metastasis. This serves as a gold-standard endpoint for assessing the long-term efficacy of anticancer therapy.
Organ Preservation Rate (OPR) | 1 month after surgery
  The proportion of patients who avoid radical surgery and retain anal function and rectal organ integrity after neoadjuvant therapy, assessed at T3 (1 month after surgery for operated patients, or 1 month after treatment plan confirmation for non-operated patients, corresponding to the technical roadmap).
Neoadjuvant Therapy Score for Rectal Cancer (NAR) | Post-neoadjuvant Therapy Efficacy Assessment Time Point (within 8-12 weeks after radiotherapy completion)
  At T2 (8-14 weeks after the end of neoadjuvant therapy), the patient's response to neoadjuvant therapy is evaluated using a standardized scoring system that integrates endoscopic findings, imaging regression, and tumor marker levels.
Quality of Life (QoL) | Baseline (T0), within 2 weeks after completion of radiotherapy (T1), 8-12 weeks after completion of radiotherapy (T2), and 4 weeks after surgery or after final treatment regimen determination (T3), through study completion, an average of 1 year
  Assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) and Colorectal Cancer-Specific Module (EORTC QLQ-CR29) to evaluate physical function, psychological status, and bowel-related quality of life. The EORTC QLQ-C30 uses a 0-100 scale where higher scores in functional domains indicate better function, and higher scores in symptom domains indicate worse symptoms. The EORTC QLQ-CR29 uses a 0-100 scale where higher scores in symptom domains indicate worse bowel/rectal symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes